CLINICAL TRIAL: NCT05510310
Title: Breast Stimulation vs. Low Dose Oxytocin Augmentation for Women With a History of One Prior Cesarean Section Scar and in Grand Multiparas
Brief Title: Breast Stimulation vs. Low Dose Oxytocin Augmentation for Labor Induction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, Director of the Mother and Fetus Unit, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0101-21-NHR
Record Dates: First submitted 2022-08-05; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Labor Onset and Length Abnormalities; Uterine Rupture; Birth; Induced
Keywords: labor induction; birth augmentation; uterine scarring; caesarian section
MeSH Terms: conditions — Uterine Rupture | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: prospective, two-arm, active-comparator, randomized, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Breast stimulation (Experimental): Breast pump for breast stimulation: The suction cup will be placed on the breast, held by the patient or a strap, alternated between nipples every 15 minutes, with a pause of 15 minutes after each 30 minutes. Suction intensity will be adjusted to the maximum tolerated by the patient while avoiding causing pain or discomfort. Treatment will be continued for a maximum of 12 hours.
  Interventions: Procedure: Breast stimulation
- Low-dose oxytocin (Active Comparator): Low-dose oxytocin will be administered intravenously, starting at a dose of 0.5-2 milliunits\minute, and increasing incrementally by 1-2 milliunites\minute every 15-40 minutes. Treatment will be continued for a maximum of 12 hours.
  Interventions: Biological: Oxytocin

INTERVENTIONS:
Procedure: Breast stimulation — By breast pump
  Arms: Breast stimulation
Biological: Oxytocin — Oxytocin will be administered intravenously and titrated
  Arms: Low-dose oxytocin

SUMMARY:
To find the preferred method of labor induction (birth augmentation) for women with a history of one prior cesarean section scar and in grandmultiparas, the difference in time interval from augmentation to delivery will be measured between breast stimulation vs. low-dose oxytocin administration in this prospective single-center randomized controlled trial.

DETAILED DESCRIPTION:
Introduction The primary cause of uterine scars is a previous cesarean. In women with a previous cesarean, the risks of maternal complications are rare and similar after a trial of labor after cesarean (TOLAC) and after an elective repeat cesarean delivery (ERCD), but the risk of uterine rupture is higher with TOLAC (0.2-0.8%)[1] . Maternal morbidity in women with previous cesareans is higher when TOLAC fails than when it leads to successful vaginal delivery[2]. Although maternal morbidity increases progressively with the number of ERCD, maternal morbidity of TOLAC decreases with the number of successful previous TOLAC[2].

Induction of labor is a common procedure undertaken whenever the benefits of prompt delivery outweigh the risks of expectant management. The goal of labor induction is to ensure the best possible outcome for mother and newborn[3].

For women after cesarean delivery labor should be induced only for medical indications[4]. Induction during TOLAC moderately increases the risk of cesarean delivery during labor, but approximately doubles the risk of uterine rupture compared with spontaneous labor in women with uterine scars[4].

Breast stimulation for inducing uterine contractions has been reported in the medical literature since the 18th century.

The American college of Obstetricians and Gynecologists (ACOG) has described nipple stimulation as a natural and inexpensive nonmedical method for inducing labor. Stimulation of the nipple by manual rolling of the nipple as well as by the breast pump has been used for performing contraction stress tests, induction or augmentation of labor and for reducing blood loss in the third stage of labor[5]. Nipple and uterine stimulation reduce the frequency of elective labor induction, the rate of relevant complications, and support normal vaginal birth by providing endogenous labor induction[6]. The mechanical uterotonic effect of breast stimulation is well recognized and described as a means of facilitating uterine contractions[7][8]. Breast stimulation can ripen the cervix in term pregnancy, seen as dilation and effacement, causing a change in Bishop score and increasing the incidence of spontaneous labor[9][10][11] A systematic review previously reported that breast stimulation for labor induction reduced the number of women who were not in labor after 72 h [12].

The success rate of breast stimulation in causing spontaneous labor varies from 45% to 84% of women undergoing induction of labor in term pregnancy[7][9][13] In a study published by Shalev et al. (1990), the effect of breast stimulation on the prostaglandin secretion was tested in 13 patients at 38-40 weeks of gestation. Uterine contractions following breast stimulation were documented in all cases. There was an increase in prostaglandin metabolite levels 10 min after breast stimulation[8]. Breast stimulation was also found to cause elevation in plasma and salivary oxytocin levels[5][14].

Oxytocin is a key hormone in childbirth, and synthetic oxytocin is widely administered to induce or speed labor. In women with a favorable cervix, combined use of amniotomy and intravenous oxytocin is generally the most effective approach[3]. A systematic review published by Uvnäs-Moberg et al. (2019) stated that oxytocin levels following infusion of synthetic oxytocin up to 10 millinuits/minute (mU/min) were similar to oxytocin levels in physiological labor[14]. Oxytocin in the circulation stimulates uterine contractions, and oxytocin released within the brain influences maternal physiology and behavior during birth.

Regarding the choice of induction using synthetic oxytocin vs. breast stimulation, a study by Mashini et al. (1987) found that a significant increase in uterine activity, measured by internal pressure catheter and quantified in Montevideo units, occurred in both treatments. [15]. The authors stated that exogenous oxytocin and intermittent nipple stimulation may not have equivalent effects on uterine contractility, since 20% of women induced by breast stimulation did not achieve adequate contraction patterns after 15 stimulation-rest cycles (a total of 110 min). Breast stimulation in this study was performed manually by the gravida by stroking the nipple using the palmar surface of the hand over the gown for two minutes followed by a five-minute rest period.

The use of breast stimulation could be recommended when oxytocin is advised to be given with caution or low doses for higher risk pregnancies. A retrospective study in 135 women by Segal et al. (1995) concluded that breast stimulation in grandmultiparas (birth number 6 and above) and in women with a previous cesarean section is efficacious and safe[13]. The results did not specify the P value of analysis between the study groups, failed to define a group of patients in whom the success rate of induction by breast stimulation significantly differed from that of other groups, and stated that "studies comparing breast stimulation with oxytocin may further define its role." Women with a history of one prior cesarean section scar or grandmultipara are deemed to have a relative contraindication to induction of labor with high-dose oxytocin for the risk of uterine rupture or overstimulation.

In this study, the researchers aim to define the preferred mode of augmentation for such cases.

Study design A prospective single-center randomized controlled trial (*Department of Obstetrics and Gynecology, Galilee Medical Center, Nahariya) Written informed consent will be obtained from all participants before randomization.

Aim: To examine the difference and finding the preferred mode of birth augmentation for women with a history of one prior cesarean section scar and in grandmultiparas. For each type of augmentation, an assessment will be made of Montevideo levels that indicate effective augmentation.

Inclusion criteria:

1. Singleton vertex gestations at or beyond 37 weeks of gestation
2. History of one prior cesarean section scar or grandmultipara (birth number 6 and above),
3. Spontaneous onset of labor or after labor induction by Foley balloon catheter
4. Determined by the obstetrics care team that augmentation was needed.
5. Augmentation will be initiated at or beyond 2.5 cm dilation, with or without ruptured membranes and uterine activity less than 3 contractions in 10 min on tocodynamometry.

Exclusion criteria:

1. History of two prior cesarean section scars
2. Younger than 18 years
3. Any contraindication for vaginal birth (placenta previa, vasa previa, cord presentation, inadequate pelvis, prior uterine rupture),
4. Fetuses in nonvertex presentation
5. fetuses with suspected life-limiting anomalies,
6. Suspected abruption or bleeding of unknown origin,
7. Women who did not agree to the enter the study.

Endpoints Primary endpoint: Time interval from augmentation to delivery Secondary endpoints: Montevideo units measured in the active first and second stage of labor, women who achieved vaginal delivery, gravida satisfaction for augmentation treatment, clinical chorioamnionitis, endometritis, postpartum hemorrhage, Apgar score 3 or less at 5 minutes, umbilical artery acidemia, neonatal intensive care unit admission, perinatal death, and severe perinatal morbidity composite Study hypothesis: A significant difference in time interval from augmentation to delivery will be measured between breast stimulation vs. low-dose oxytocin augmentation.

Methods Pregnant women satisfying the enrollment criteria and providing informed consent will be randomly selected for augmentation by breast pump for breast stimulation (as described below) or by an IV low-dose oxytocin course (starting dose 0.5-2 mU/min and increasing the dose incrementally by 1-2mU\min every 15-40 min). Both augmentation treatments will be continued for a maximum of 12 hours.

Breast pump for breast stimulation: The suction cup will be placed on the breast, held by the patient or a strap, alternated between nipples every 15 minutes, with a pause of 15 minutes after each 30 minutes. Suction intensity will be adjusted to the maximum tolerated by the patient while avoiding pain or discomfort.

Augmentation will be initiated at or beyond 2.5 cm dilation, minimum Bishop score of 6, with or without ruptured membranes, uterine activity less than 3 contractions in 10 minutes on tocodynamometry.

Uterine activity will be measured by an intrauterine pressure catheter that will be placed after spontaneous or artificial rupture of membranes at or beyond 2.5 cm dilation.

The augmentation will be adjusted if uterine overstimulation occurs (above 5 contractions in 10 minutes).

The augmentation will be stopped if uterine overstimulation persists, if non-reassuring fetal heart rate tracing occurs, discontinuing the treatment is deemed necessary, or following the patient's choice.

In cases with unruptured membranes, induction will be carried out for various medical and obstetric indications (post-term, oligohydramnios, etc.) after cervical ripening with catheter balloon if needed.

In cases of ruptured membranes, labor will be induced if it did not ensue spontaneously within 24 hours of spontaneous rupture of membranes.

Spontaneous onset of labor is defined as the presence of at least 6 spontaneous contractions per hour on tocodynamometry with either spontaneous rupture of membranes, or intact membranes with at least 3 cm of cervical dilation or 80% cervical effacement.

In addition, the following data will be collected: gravida age, ethnicity, gestational age at admission and birth, indication for induction, reason for birth by cesarean section, background diseases, and diseases complicating pregnancy.

Statistical analysis A sample size of 100 patients in each group was calculated using data from research by Mashini et al. (1987), which published time from augmentation to delivery and uterine activity measured in Montevideo units after induction by nipple stimulation vs. oxytocin infusion [15].

Power analysis was calculated in order to compare time from augmentation to delivery between breast stimulation vs. low-dose oxytocin augmentation.

A difference of at least 2 units between the groups (for example, 9.5±4.3 vs. 7.5±2.6, respectively) is anticipated.

Based on independent t-test 2-side hypothesis testing with alpha=5% and 70 women in each group, the power is 91%.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton vertex gestations at or beyond 37 weeks of gestation
2. History of one prior cesarean section scar or grandmultipara (birth number 6 and above),
3. Spontaneous onset of labor or after labor induction by Foley balloon catheter, eligible for this trial
4. Determined by the obstetrics care team that augmentation was needed.
5. Augmentation will be initiated at or beyond 2.5 cm dilation, with or without ruptured membranes and uterine activity less than 3 contractions in 10 minutes on tocodynamometry.

Exclusion Criteria:

1. History of two prior cesarean section scars,
2. Younger than 18 years,
3. Any contraindication for vaginal birth (placenta previa, vasa previa, cord presentation, inadequate pelvis, prior uterine rupture),
4. Fetuses in nonvertex presentation
5. Fetuses with suspected life-limiting anomalies,
6. Suspected abruption or bleeding of unknown origin,
7. Women who did not agree to the enter the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Time interval from augmentation of labor to delivery | up to 48 hours

SECONDARY OUTCOMES:
Montevideo units in each group | active first and second stage of labor (up to 48 hours)
rate of women who achieved vaginal delivery | during labor (48 hours)
Endometritis | during one week postpartum
  fever abdominal pain
Postpartum hemorrhage | during the first 24 hours after labor
Apgar score 3 or less at 5 minutes | during the first 5 minutes postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Maya Wolf, MD, Principal Investigator — Galilee Medical Center
Locations (1):
- Galil Medical Center, Nahariya, Israel

REFERENCES:
- [Background] Sentilhes L, Vayssiere C, Beucher G, Deneux-Tharaux C, Deruelle P, Diemunsch P, Gallot D, Haumonte JB, Heimann S, Kayem G, Lopez E, Parant O, Schmitz T, Sellier Y, Rozenberg P, d'Ercole C. Delivery for women with a previous cesarean: guidelines for clinical practice from the French College of Gynecologists and Obstetricians (CNGOF). Eur J Obstet Gynecol Reprod Biol. 2013 Sep;170(1):25-32. doi: 10.1016/j.ejogrb.2013.05.015. Epub 2013 Jun 28. PMID 23810846
- [Background] Beucher G, Dolley P, Levy-Thissier S, Florian A, Dreyfus M. [Maternal benefits and risks of trial of labor versus elective repeat caesarean delivery in women with a previous caesarean delivery]. J Gynecol Obstet Biol Reprod (Paris). 2012 Dec;41(8):708-26. doi: 10.1016/j.jgyn.2012.09.028. Epub 2012 Nov 14. French. PMID 23159201
- [Background] Penfield CA, Wing DA. Labor Induction Techniques: Which Is the Best? Obstet Gynecol Clin North Am. 2017 Dec;44(4):567-582. doi: 10.1016/j.ogc.2017.08.011. PMID 29078939
- [Background] Deruelle P, Lepage J, Depret S, Clouqueur E. [Induction of labor and intrapartum management for women with uterine scar]. J Gynecol Obstet Biol Reprod (Paris). 2012 Dec;41(8):788-802. doi: 10.1016/j.jgyn.2012.09.030. Epub 2012 Nov 9. French. PMID 23142358
- [Background] Christensson K, Nilsson BA, Stock S, Matthiesen AS, Uvnas-Moberg K. Effect of nipple stimulation on uterine activity and on plasma levels of oxytocin in full term, healthy, pregnant women. Acta Obstet Gynecol Scand. 1989;68(3):205-10. doi: 10.3109/00016348909020990. PMID 2618602
- [Background] Demirel G, Guler H. The Effect of Uterine and Nipple Stimulation on Induction With Oxytocin and the Labor Process. Worldviews Evid Based Nurs. 2015 Oct;12(5):273-80. doi: 10.1111/wvn.12116. PMID 26444882
- [Background] Jhirad A, Vago T. Induction of labor by breast stimulation. Obstet Gynecol. 1973 Mar;41(3):347-50. No abstract available. PMID 4688251
- [Background] Shalev E, Weiner E, Tzabari A, Engelhard J, Zuckerman H, Shalev J, Serr DM. Breast stimulation in late pregnancy. Effect on prostaglandin secretion. Gynecol Obstet Invest. 1990;29(2):125-7. doi: 10.1159/000293317. PMID 2335311
- [Background] Elliott JP, Flaherty JF. The use of breast stimulation to ripen the cervix in term pregnancies. Am J Obstet Gynecol. 1983 Mar 1;145(5):553-6. doi: 10.1016/0002-9378(83)91194-8. PMID 6338721
- [Background] Kavanagh J, Kelly AJ, Thomas J. Breast stimulation for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD003392. doi: 10.1002/14651858.CD003392.pub2. PMID 16034897
- [Background] Singh N, Tripathi R, Mala YM, Yedla N. Breast stimulation in low-risk primigravidas at term: does it aid in spontaneous onset of labour and vaginal delivery? A pilot study. Biomed Res Int. 2014;2014:695037. doi: 10.1155/2014/695037. Epub 2014 Nov 27. PMID 25525601
- [Background] Kavanagh J, Kelly AJ, Thomas J. Breast stimulation for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2001;(4):CD003392. doi: 10.1002/14651858.CD003392. PMID 11687199
- [Background] Segal S, Gemer O, Zohav E, Siani M, Sassoon E. Evaluation of breast stimulation for induction of labor in women with a prior cesarean section and in grandmultiparas. Acta Obstet Gynecol Scand. 1995 Jan;74(1):40-1. doi: 10.3109/00016349509009941. PMID 7856430
- [Background] Uvnas-Moberg K, Ekstrom-Bergstrom A, Berg M, Buckley S, Pajalic Z, Hadjigeorgiou E, Kotlowska A, Lengler L, Kielbratowska B, Leon-Larios F, Magistretti CM, Downe S, Lindstrom B, Dencker A. Maternal plasma levels of oxytocin during physiological childbirth - a systematic review with implications for uterine contractions and central actions of oxytocin. BMC Pregnancy Childbirth. 2019 Aug 9;19(1):285. doi: 10.1186/s12884-019-2365-9. PMID 31399062
- [Background] Mashini IS, Devoe LD, McKenzie JS, Hadi HA, Sherline DM. Comparison of uterine activity induced by nipple stimulation and oxytocin. Obstet Gynecol. 1987 Jan;69(1):74-8. PMID 3796923